CLINICAL TRIAL: NCT06135038
Title: Does Shoulder Injection in Patients With Chronic Shoulder Pain Contribute to Physiotherapy?
Brief Title: Injection in Patients With Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Kagan Ozkuk, Assoc. Prof., Uşak University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Physical Medicine+injection
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Shoulder Pain
Keywords: chronic shoulder pain; shoulder injection; suprascapular nerve block; physiotherapy
MeSH Terms: interventions — Physical Therapy Modalities; Transcutaneous Electric Nerve Stimulation; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprascapular nerve block with physical therapy (Active Comparator): Suprascapular Nerve Block was applied to Group I before physical therapy program.
  After the nerve block, a physical therapy program including standard procedure was applied to the patients in Group 1.
  Interventions: Other: Suprascapular nerve block with physical therapy
- Only physical therapy (Active Comparator): Patients in group 2 were applied only a physical therapy program that included the same standard procedure as group 1.
  Interventions: Other: Group 2 Physical therapy

INTERVENTIONS:
Other: Suprascapular nerve block with physical therapy — Suprascapular nerve block was applied to the relevant shoulder area of all patients before treatment. Afterwards, a physical therapy program (5 days a week for 3 weeks, a total of 15 sessions) was applied, including 20 minutes of hot pack at 60°C, 20 minutes of conventional TENS at 80 Hz and US at 3 MHz frequency and 1.5 watt/cm2 intensity.
  After physical therapy, all the participants received therapeutic exercise program (3 sets of 10 reps with 3- minute intervals between the sets) consisting of active-assisted ROM, passive stretching and Codman exercises for their shoulder joint for 30 minutes in accompany with a physiotherapist.
  Other Names: Transcutaneous Electrical Nerve Stimulation (TENS); Hot Pack; Ultrasound(US) Therapy; Therapeutic Exercise Program
  Arms: Suprascapular nerve block with physical therapy
Other: Group 2 Physical therapy — A physical therapy program (5 days a week for 3 weeks, a total of 15 sessions), including a hot pack at 60 ° C for 20 minutes, conventional TENS at 80 Hz for 20 minutes and US at 3 MHz frequency and an intensity of 1.5 watts / cm2, was applied to the relevant shoulder area of all patients.
  After physical therapy, all the participants received therapeutic exercise program (3 sets of 10 reps with 3- minute intervals between the sets) consisting of active-assisted ROM, passive stretching and Codman exercises for their shoulder joint for 30 minutes in accompany with a physiotherapist.
  Other Names: Transcutaneous Electrical Nerve Stimulation (TENS); Hot Pack; Ultrasound(US) Therapy; Therapeutic Exercise Program
  Arms: Only physical therapy

SUMMARY:
Background: Chronic shoulder pain (CSP) is a musculoskeletal disease characterized by pain lasting more than 3 months.

Purpose: This study aimed to determine whether pre-treatment injection in CSP treatment contributes to pain, functionality and quality of life.

Methods: A total of 110 patients who met the inclusion criteria of the study were divided into 2 groups (55 patients in each group).

A standard 15-session physical therapy program (hot pack, transcutaneous electric nerve stimulation(TENS), US and therapeutic exercises) was applied to all patients in both groups. Suprascapular Nerve Block was applied to Group I before treatment.

Assessments were made using VAS-Pain, Shoulder Pain and Disability Index (SPADI) and The Nottingham Health Profile (NHP) before and at the end of the treatment and in the posttreatment 3th months.

DETAILED DESCRIPTION:
INTRODUCTION Chronic pain is a common condition, affecting 20% of people worldwide and accounting for 15% to 20% of doctor visits. One of the most common causes of chronic pain and disability in the world is musculoskeletal system diseases. Pain and limitations in daily living activities and psychological problems that develop due to pain negatively affect the quality of life of patients.

Shoulder pain is the third most common musculoskeletal system disease that causes pain and loss of function. Shoulder pain is characterized by chronicity and high recurrence rates due to its anatomy and joint structure.

Chronic and frequently recurring shoulder pain can cause loss of function and not only affects the individual's entire life, but also becomes a socio-economic problem with the financial burden it brings.

There are many pharmacological or non-pharmacological treatment approaches in the treatment of pain. Many physical therapy methods are used in combination for chronic shoulder pain (e.g. Hotpack, TENS, ultrasound, exercise, etc.). Alternative treatments and their combinations are gaining importance today in painful shoulder problems that are difficult to treat with physiotherapy due to their anatomical and functional structure.

This study aimed to determine whether pre-treatment injection in CSP treatment contributes to pain, functionality and quality of life.

METHODS The study was designed as a prospective, randomized, controlled, and single-blind study. A total of 110 patients who were admitted to the physical therapy and rehabilitation outpatient clinic with pain and movement restriction in their shoulder and who signed the patient information consent form were included in the study.

A total of 110 patients who met the inclusion criteria of the study were divided into 2 groups (55 patients in each group) with simple randomization method by using a table of random numbers created on the computer. The researchers who made the assessment measurements were unaware of which patient was in which group. Statistical analysis of the results was performed by a biostatistician who had no information about the therapies the patient groups received.

All the patients included in the study received a total of 15 sessions of physical therapy program 5 times a week for 3 weeks. All the patients received hot pack at 60°C for 20 minutes and conventional TENS at 80 Hz for 20 minutes and US at 3 megahertz frequency, and 1.5watt/cm2 intensity for their involved shoulder. After physical therapy, all the participants received therapeutic exercise program (3 sets of 10 reps with 3- minute intervals between the sets) consisting of active-assisted range of motion (ROM), passive stretching and Codman exercises for their shoulder joint for 30 minutes in accompany with a physiotherapist. Suprascapular Nerve Block was applied to Group I before treatment. The patients were assessed with the measurements of visual analogue scale (VAS)-pain, Shoulder Pain and Disability Index (SPADI) and The Nottingham Health Profile (NHP) before and immediately after the intervention and at 12 weeks after the end of the intervention (approximately week 15).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Having pain lasting longer than 3 months,
* Full range of joint motion
* Patients with shoulder pain due to biceps tendinitis, impingement syndrome, rotator cuff diseases (tendinosis, calcific tendonitis, etc.)

Exclusion Criteria:

* Inflammatory rheumatic disease (rheumatoid arthritis, ankylosing spondylitis, etc.),
* Full thickness rotator cuff tear
* Glenohumeral disorders (arthritis, osteoarthritis, osteonecrosis, glenohumeral instability)
* Regional disorders (cervical radiculopathy, brachial neuritis, entrapment neuropathies, reflex sympathetic dystrophy, neoplasms, etc.)
* Diagnosed with metabolic syndrome, diabetes mellitus (DM), hypertension (HT)
* Having a diagnosed neuro-psychiatric problem,
* Undergoing malignancy treatment,
* Having a bleeding disease,
* Having an infectious disease with fever,
* Who have undergone surgery on the shoulder,
* Patients who received physical therapy in the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS)-pain | Outcome measure evaluated; 1. Before the intervention, 2. Immediately after the intervention, 3. At 12 weeks after the end of the intervention (approximately week 15)
  Visual analogue scale (VAS) is one of the frequent methods used in the identification of the severity of pain. It is formed by 100 mm vertical and horizontal lines. The distance between the lowest VAS score and the mark of the patient was measured as mm (0-100) and the numerical value of the pain severity was determined .
Shoulder Pain and Disability Index (SPADI) | Outcome measure evaluated; 1. Before the intervention, 2. Immediately after the intervention, 3. At 12 weeks after the end of the intervention (approximately week 15)
  The shoulder Pain and Disability Index was developed to evaluate pain and disability . It consists of 2 subscales, consisting of a total of 13 items (5 items for pain, 8 items for disability) numerically rated from 0 to 10. The total score ranges from 0 to 100. Higher scores represent increased pain and impaired shoulder function.
The Nottingham Health Profile (NHP) | Outcome measure evaluated; 1. Before the intervention 2. Immediately after the intervention, 3. At 12 weeks after the end of the intervention (approximately week 15)
  The Nottingham Health Profileis a general quality of life questionnaire measuring self-perceived health problems and the effects of these problems on normal daily activities. The questionnaire consists of 38 questions and six domains. For each domain, "0" represents the best state of health and "100" the worst state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Kağan Özkuk, Study Director — Uşak University
Locations (1):
- UsakU, Merkez, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No